CLINICAL TRIAL: NCT02678208
Title: The Effect of Tranexamic Acid on Uterine Blood Flow After Vaginal Delivery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TBBH
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Postpartum Hemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic acid (Active Comparator): received tranexamic acid containing 1 g/10mL tranexamic acid diluted with 20 mL of 5% glucose over a 5 minute period
  Interventions: Drug: Tranexamic Acid; Drug: 5% glucose
- placebo (Other): received 30 mL of 5% glucose over the same period of time.
  Interventions: Drug: 5% glucose

INTERVENTIONS:
Drug: Tranexamic Acid
  Arms: Tranexamic acid
Drug: 5% glucose

SUMMARY:
Postpartum hemorrhage is the most common cause of maternal death across the world, responsible for more than 25% of maternal deaths annually. Although effective tools for prevention and treatment of are available, most are not feasible or practical for use in the developing world where many births still occur at home with untrained birth attendants . primary postpartum hemorrhage is excessive bleeding from or in the genital tract within 24 hours of delivery of the fetus which affects the general condition.

Postpartum hemorrhage is responsible for around 25% of maternal mortality worldwide , reaching as high as 60% in some countries. Postpartum hemorrhage can also be a cause of long-term severe morbidity, and approximately 12% of women who survive postpartum hemorrhagewill have severe anemia.

Tranexamic acid is an antifibrinolytic compound which is a potent competitive inhibitor of the activation of plasminogen to plasmin. At much higher concentrations it is a non-competitive inhibitor of plasmin. The inhibitory effect of tranexamic acid in plasminogen activation by urokinase has been reported to be 6-100 times and by streptokinase 6-40 times greater than that of aminocaproic acid.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women (37-42 weeks),
* with spontaneous labor
* Women who were expected to normal vaginal birth.
* women with a live fetus.

Exclusion Criteria:

* multiple gestations
* polyhydramnios
* macrocosmic baby
* grand multipara
* women with hypertensive disorders
* previous history of postpartum hemorrhage
* abnormal placentation (placenta previa or placental abruption)
* history of any uterine scarring (including cesarean section)
* history of blood/liver/renal/heart diseases.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The changes in Doppler indices of uterine artery after use of tranexamic acid | 6 months
The changes in Doppler indices of intramyometrial blood vessels after use of tranexamic acid | 6 months
The changes in Doppler indices of subendomterial blood vessels after use of tranexamic acid | 6 month

SECONDARY OUTCOMES:
The volume of blood loss after delivery (mL) | 6 months
Number of patients needed for blood transfusion | 6 months
The hematocrit values (%) | 6 months
The hemoglobin concentration | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes